CLINICAL TRIAL: NCT04495283
Title: A Phase 2, Randomized, Double-Blind, Placebo- and Comparator-Controlled Trial to Evaluate the Safety and Efficacy of Combination of Pregabalin and Acetaminophen Compared to Acetaminophen and Placebo in Subjects Undergoing Bunionectomy
Brief Title: A Phase 2 Study to Evaluate Pregabalin and Acetaminophen Compared to Acetaminophen and Placebo in Subjects Undergoing Bunionectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nevakar, Inc. (Industry)
Collaborators: Nevakar Injectables, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CP-NVK009-0005
Record Dates: First submitted 2020-07-27; First posted 2020-07-31 (Actual); Results first posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin; Prostaglandins B; Acetaminophen

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator
Masking Description: Up to 80 subjects will be randomized (32 in each active treatment group, 16 placebo).
  Eligible subjects will be randomized on Day 1 in a 2:2:1 ratio to receive either a combination of PGB and APAP administered (Group A), APAP (Group B), or placebo (Group C).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PGB and APAP (Group A) (Experimental): Group A receives PGB plus APAP prior to surgery and placebo 1 post-surgery.
  Interventions: Drug: Pregabalin; Drug: Acetaminophen
- APAP (Group B) (Experimental): Group B receives placebo 2 prior to surgery and APAP post-surgery.
  Interventions: Drug: Acetaminophen; Other: Placebo 2
- Placebo (Group C). (Experimental): Group C receives placebo 1 prior to surgery and placebo 2 post-surgery.
  Interventions: Other: Placebo 1; Other: Placebo 2

INTERVENTIONS:
Drug: Pregabalin — Pregabalin is a structural derivative of the inhibitory neurotransmitter gamma aminobutyric acid with anticonvulsant, anxiolytic and sleep-modulating properties.
  Other Names: PGB
  Arms: PGB and APAP (Group A)
Drug: Acetaminophen — Acetaminophen is a non-salicylate antipyretic and non-opioid analgesic agent.
  Other Names: APAP
  Arms: APAP (Group B); PGB and APAP (Group A)
Other: Placebo 1 — Placebo for APAP
  Arms: Placebo (Group C).
Other: Placebo 2 — Placebo for combination
  Arms: APAP (Group B); Placebo (Group C).

SUMMARY:
A Phase 2, Randomized, Double-Blind, Placebo- and Comparator-Controlled Trial to Evaluate the Safety and Efficacy of Combination Pregabalin and Acetaminophen Compared to Acetaminophen and Placebo in Subjects Undergoing Bunionectomy

DETAILED DESCRIPTION:
A Phase 2, Randomized, Double-Blind, Placebo- and Comparator-Controlled Trial to Evaluate the Safety and Efficacy of Combination Pregabalin and Acetaminophen Compared to Acetaminophen and Placebo in Subjects Undergoing Bunionectomy

Up to 80 subjects will be randomized (32 in each active treatment group, 16 placebo).

To evaluate the efficacy of combination pregabalin (PGB) and acetaminophen (APAP) administered vs. placebo for pain control in subjects undergoing bunionectomy.

The placebo will be the saline solution.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent by signing the informed consent form (ICF) approved by the Institutional Review Board (IRB);
* Be male or female aged 18-65 years;
* Be scheduled to undergo unilateral first metatarsal bunionectomy;
* Be in good health and capable of undergoing a bunionectomy under anesthesia as described in the study surgical and anesthetic protocol;
* Weigh between 50 and 100 kg (body mass index [BMI] <32 kg/m2);
* Have no additional planned surgeries other than bunionectomy during the course of the study;
* Have negative urine drug screen for drugs indicative of illicit drug use (unless results can be explained by a current prescription or acceptable over-the-counter medication at screening as determined by the investigator) and no detectable results on the alcohol test (breath or saliva) indicative of alcohol abuse at screening, and/or prior to surgery (may be repeated if the Investigator suspects a false-positive result). Note: For those subjects who test positive for tetrahydrocannabinol (THC), if they are willing to abstain from use or consumption of THC-containing products from screening through end of the subject's participation in the study, they may be allowed to participate in the study.
* Biological female subjects must be non-lactating, sterile (bilateral tubal ligation, bilateral salpingectomy, or hysterectomy), post-menopausal for at least 2 years, have a partner that is sterile, be abstinent, use a highly effective double- contraception method (hormonal protection is insufficient), or use an FDA-approved contraceptive for greater than 2 months prior to the screening visit and commit to an acceptable form of birth control for the duration of the study and for 30 days after completion of the study;
* Be willing and able to complete the study procedures and pain scales and communicate meaningfully in English with study personnel.

Exclusion Criteria:

* Have a medical condition or history that in the Investigator's opinion could adversely impact the subject's participation or safety or the conduct of the study, or interfere with the pain assessments, including the following:

  1. Serious breathing difficulties or respiratory risk factors (including use of opioid pain medicines and other drugs that depress the central nervous system), and conditions such as chronic obstructive pulmonary disease that reduce lung function.
  2. Hypertension (uncontrolled), cardiovascular disease, or history of cerebrovascular events. Hypertension must be controlled without known end organ damage.
  3. Concurrent painful conditions that may require analgesic treatment during the study period.
  4. History of significantly reduced hepatic or renal function, angle closure glaucoma, or convulsive disorder.
  5. Recent history of urinary retention.
  6. Opioid tolerant, i.e., the subject is currently taking or has taken a chronic opioid at a dose greater than or equal to 20 mg morphine milligram equivalents (MME) per day (more than 30 consecutive days of daily use) for pain in the 2 months prior to surgery.
  7. Active cutaneous disease, or other disease, at the surgical site.
  8. Peripheral vascular disease, sickle cell disease, vascular grafts, or vasospastic disorders.
  9. Known bleeding disorder or is taking agents affecting coagulation preoperatively.

     Deep venous thrombosis (DVT) prophylaxis of the surgeon's choice is permitted postoperatively.
  10. Diabetes mellitus (uncontrolled). Diabetes mellitus must be controlled without known end organ damage.
  11. History of malignancy in the past 2 years with the exception of squamous cell carcinoma or basal cell carcinoma.
  12. Prior bunionectomy on the index foot or other foot surgery on the index foot that could impact the surgery or data collection endpoints.
* Use of disallowed medications including the following:

  1. Pain medication (opioids, NSAIDs, cyclooxygenase (COX)-2 inhibitors, tramadol, ketamine, clonidine, gabapentin, pregabalin, or cannabinoids) within 2 days prior to Day 1.
  2. Central nervous system (CNS) active drugs such as benzodiazepines, tricyclic antidepressants, serotonin and norepinephrine reuptake inhibitors (SNRIs), or selective serotonin reuptake inhibitors (SSRIs) for pain within seven days prior to Day 1. These drugs are permitted for non-pain indications if the dose has been stable for at least 30 days prior to Day 1 and is planned to remain stable throughout the study. The use of lorazepam and other sleep medications, except those containing analgesic properties, is permitted.
  3. Use of parenteral or oral corticosteroid(s) within 14 days prior to Day 1.
  4. Antihypertensive agent or diabetic regimen at a dose that has not been stable for at least 30 days, or which is not expected to remain stable throughout the study.
  5. Digoxin, warfarin (see exception below), lithium, theophylline preparations, aminoglycosides, and all antiarrhythmics except beta-blockers, and use of anticonvulsants except benzodiazepines within 7 days prior to Day 1 and throughout the study.
* Use of warfarin is allowed, at the investigator's discretion, for DVT prophylaxis after the surgery.
* Significant history of allergic reactions or known intolerance to pregabalin or any gabapentinoid, to APAP, to any rescue medication used in the study, or any medication used in the surgical and anesthetic protocol.
* Female subjects (biological females only) who are pregnant or lactating, who plan to get pregnant, or who have a positive serum pregnancy test at Screening or a positive urine pregnancy test at either Day -1 or Day 1 prior to surgery.
* Participated in another clinical trial within 30 days, or previously participated in a clinical study with a similar investigational product.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Lotus Clinical Resarch,LLC, Pasadena, California
  - Lotus HD Research, Bellaire, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 28 July 2020 till 26 Oct 2020 across the sites.
Pre-assignment Details: Subjects underwent a Screening Visit (Day -42 to Day -2) and were required to sign an informed consent form (ICF) before undertaking any study-specific procedures or assessments. Pre-operative assessments were conducted within 24 hours prior to surgery (on either Day -1 or Day 1 prior to surgery.
Groups:
- PGB and APAP (Group A): Group A receives pregabalin (PGB) plus acetaminophen (APAP) prior to surgery and placebo 1 post-surgery.
Period: Overall Study
Arm/Group | PGB and APAP (Group A) | APAP (Group B) | Placebo (Group C).
Started | 35 | 35 | 17
Completed | 34 | 34 | 14
Not Completed | 1 | 1 | 3
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Other | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all subjects who received any amount of study drug (APAP + PGB, APAP, or placebo), whether or not they were prematurely withdrawn from the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | PGB and APAP (Group A) | APAP (Group B) | Placebo (Group C). | Total
Number analyzed (Participants) | 35 | 35 | 17 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (13.33) | 42.1 (11.68) | 43.3 (11.98) | 43.0 (12.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 31 | 17 | 73
  Male | 10 | 4 | 0 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 12 | 7 | 28
  Not Hispanic or Latino | 26 | 23 | 10 | 59
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 1 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 7 | 4 | 18
  White | 24 | 26 | 12 | 62
  More than one race | 2 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.03 (3.213) | 26.55 (3.471) | 26.05 (3.406) | 26.24 (3.326)

OUTCOME MEASURES:

1. Primary Outcome: Summed Pain Intensity (SPI) Between Group A and Group C
Description: Pain Intensity using a pain rating of 0-10 on the Numerical Rating Scale (NRS), with a score between 0-10 (0= no pain; 10 = worst imaginable pain). Summed Pain Intensity (SPI0-48) was calculated using the trapezoidal method as the area under the curve (AUC) of pain intensity as measured using the NRS through various time intervals up to 48 hours. For SPI0-48 calculation, all available NRS pain intensity scores (scheduled pain intensity, unscheduled pain intensity and pre-rescue pain intensity) from 0 to 48 hours, including any imputed values, was used in the calculation. Hour 0 was defined as the time of the end of surgery. SPI0-48 was calculated using the formula: Sum (1/2 (SPIi + SPIi+1)*Δt), where Δt was the time difference between Time i and Time (i+1). The represented values are sum of pain intensity scores at various time points. This outcome was compared between a combination of PGB and APAP (Group A) and placebo (Group C) from Hour 0 to Hour 48 (SPI0-48)
Time Frame: 0 to 48 hours
Population: The Full Analysis Set (FAS) included all randomized subjects who received at least one dose of study drug. Subjects were analyzed according to the treatment group to which they were randomized.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | PGB and APAP (Group A) | Placebo (Group C).
Number analyzed (Participants) | 35 | 17
score on a scale | 153.08 (15.238) | 267.51 (21.864)
Statistical Analysis 1: Comparison: PGB and APAP (Group A) vs Placebo (Group C); Test type: Superiority; p < 0.001, ANOVA; LS Mean Difference = -114.43, 90% CI 1-sided [upper limit -80.01], Standard Error of Mean 26.650

2. Secondary Outcome: Summed Pain Intensity (SPI) Compared Between Group A and Group B
Description: Pain Intensity using a pain rating of 0-10 on the Numerical Rating Scale (NRS), with a score between 0-10 (0= no pain; 10 = worst imaginable pain). Summed Pain Intensity (SPI0-48) -was calculated using the trapezoidal method as the area under the curve (AUC) of pain intensity as measured using the NRS through various time intervals up to 48 hours. For SPI0-48 calculation, all available NRS pain intensity scores (scheduled pain intensity, unscheduled pain intensity and pre-rescue pain intensity) from 0 to 48 hours, including any imputed values, were used in the calculation. Hour 0 was defined as the time of the end of surgery. SPI0-48 was calculated using the formula: SUM (1/2 (SPIi + SPIi+1)*Δt), where Δt was the time difference between Time i and Time (i+1). The represented values are sum of pain intensity scores at various time points. This outcome was compared between a combination of PGB and APAP (Group A) and APAP alone (Group B) from Hour 0 to Hour 48 (SPI0-48)
Time Frame: 0 to 48 hours
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | PGB and APAP (Group A) | APAP (Group B)
Number analyzed (Participants) | 35 | 35
score on a scale | 153.08 (15.238) | 223.24 (5.238)
Statistical Analysis 1: Comparison: PGB and APAP (Group A) vs APAP (Group B); Test type: Superiority; p < 0.001, ANOVA; LS Mean Difference = -70.16, 90% CI 1-sided [upper limit -42.32], Standard Error of Mean 21.549

3. Secondary Outcome: Summed Pain Intensity (SPI) Assessed by Numeric Rating Scale From Hour 0 to Hour 12 (SPI0-12), Hour 12 to Hour 24 (SPI12-24), and Hour 24 to Hour 48 (SPI24-48).
Description: Pain Intensity was determined using a pain rating of 0-10 on the NRS, with a score between 0-10 (0= no pain; 10 = worst imaginable pain). SPI were calculated using the trapezoidal method as the AUC of pain intensity as measured using the NRS through various time intervals at 0-12, 12-24 and 24-48 hours. For specific time interval SPI calculation, all available NRS pain intensity scores (scheduled pain intensity, unscheduled pain intensity and pre-rescue pain intensity) in the respective time interval, including any imputed values, were used in the calculation. Hour 0 was defined as the time of the end of surgery. SPI at various time intervals were calculated using the formula: SUM (1/2 (SPIi + SPIi+1)*Δt), where Δt was the time difference between Time i and Time (i+1). The represented values are sum of pain intensity scores at respective time interval (0-12, 12-24 and 24-48 hours). This outcome was compared between a combination of PGB and APAP, APAP alone, and placebo.
Time Frame: 0, 12, 24, 48 hours
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | PGB and APAP (Group A) | APAP (Group B) | Placebo (Group C).
Number analyzed (Participants) | 35 | 35 | 17
score on a scale
  SPI 0-12 | 33.09 (3.728) | 49.09 (3.728) | 58.89 (5.349)
  SPI 12-24 | 50.92 (5.082) | 69.35 (5.082) | 88.95 (7.292)
  SPI 24-48 | 126.83 (13.128) | 184.33 (13.128) | 221.58 (18.837)

4. Secondary Outcome: Summed Pain Intensity (SPI) Assessed by Numeric Rating Scale Over Time
Description: Pain Intensity was determined using a pain rating of 0-10 on the NRS, with a score between 0-10 (0= no pain; 10 = worst imaginable pain). SPI were calculated using the trapezoidal method as the AUC of pain intensity as measured using the NRS through various time intervals from 0 hour till each time point at 1, 2, 4, 6, 8, 10 ,12, 14, 16, 18, 20, 24, 28, 32, 36, 40, 44, and 48 hours. For specific time interval SPI calculation, all available NRS pain intensity scores (scheduled pain intensity, unscheduled pain intensity and pre-rescue pain intensity) in the respective time interval, including any imputed values, were used in the calculation. Hour 0 was defined as the time of the end of surgery. SPI at various time intervals were calculated using the formula: SUM (1/2 (SPIi + SPIi+1)*Δt), where Δt was the time difference between Time i and Time (i+1). The represented values are sum of pain intensity scores at respective time intervals.
Time Frame: 0, 1, 2, 4, 6, 8, 10 ,12, 14, 16, 18, 20, 24, 28, 32, 36, 40, 44, and 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PGB and APAP (Group A) | APAP (Group B) | Placebo (Group C).
Number analyzed (Participants) | 35 | 35 | 17
score on a scale
  SPI 0-1 | 0.26 (0.509) | 0.73 (0.870) | 0.45 (0.951)
  SPI 0-2 | 1.26 (1.591) | 2.39 (2.539) | 2.16 (2.560)
  SPI 0-4 | 5.63 (5.120) | 8.02 (6.703) | 9.62 (6.196)
  SPI 0-6 | 12.68 (9.650) | 17.09 (10.606) | 20.71 (10.368)
  SPI 0-8 | 20.00 (14.211) | 28.09 (14.266) | 33.64 (14.203)
  SPI 0-10 | 26.25 (18.413) | 38.71 (18.140) | 45.95 (18.510)
  SPI 0-12 | 33.09 (22.725) | 49.09 (21.692) | 58.89 (21.362)
  SPI 0-14 | 41.12 (27.035) | 58.62 (25.009) | 72.17 (24.820)
  SPI 0-16 | 49.08 (30.480) | 67.98 (27.401) | 84.46 (27.487)
  SPI 0-18 | 55.84 (33.985) | 78.49 (31.847) | 97.57 (32.420)
  SPI 0-20 | 61.49 (36.259) | 86.24 (35.453) | 108.32 (37.011)
  SPI 0-24 | 77.17 (43.864) | 108.25 (43.928) | 134.91 (42.035)
  SPI 0-28 | 88.94 (50.680) | 128.83 (52.561) | 158.01 (45.579)
  SPI 0-32 | 100.85 (56.483) | 148.93 (59.923) | 180.50 (54.648)
  SPI 0-36 | 114.43 (63.776) | 169.44 (67.178) | 203.32 (64.342)
  SPI 0-40 | 126.45 (69.998) | 186.70 (73.308) | 224.78 (72.951)
  SPI 0-44 | 139.54 (78.396) | 199.95 (78.945) | 246.09 (84.178)
  SPI 0-48 | 153.08 (87.398) | 223.24 (91.581) | 267.51 (92.791)

5. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events (TRAE)
Description: A TRAE is defined as a treatment-emergent adverse event (TEAE) that was classified by the investigator as related to study drug. The number of participants with TRAE were reported
Time Frame: 7 days
Population: The Safety Analysis Set included all subjects who received any amount of study drug (APAP + PGB, APAP, or placebo), whether or not they were prematurely withdrawn from the study. The Safety Analysis Set was used for the summaries and listings of all safety assessments. Subjects were analyzed according to treatment received
Measure: Number; unit: participants
Arm/Group | PGB and APAP (Group A) | APAP (Group B) | Placebo (Group C).
Number analyzed (Participants) | 35 | 35 | 17
participants | 22 | 9 | 7

6. Secondary Outcome: Percentage of Participants Who Were Opioid Free Over Time
Description: Percentages of participants who did not take opioid (rescue medication) over time.
Time Frame: 12 to 48 hours
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | PGB and APAP (Group A) | APAP (Group B) | Placebo (Group C).
Number analyzed (Participants) | 35 | 35 | 17
percentage of participants
  During 12-24 Hours | 65.7 | 45.7 | 35.3
  During 12-48 Hours | 48.6 | 28.6 | 29.4

7. Secondary Outcome: Total Consumption of Opioid Rescue Medication Through 24 Hours and 48 Hours
Description: The total consumption of opioid rescue analgesia through 24 hours and through 48 hours was reported
Time Frame: 24 hours and 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: oral morphine equivalents
Arm/Group | PGB and APAP (Group A) | APAP (Group B) | Placebo (Group C).
Number analyzed (Participants) | 35 | 35 | 17
oral morphine equivalents
  Consumption of Rescue Medication through 24 hours | 9.86 (14.134) | 19.24 (17.019) | 28.88 (20.981)
  Consumption of Rescue Medication through 48 hours | 17.36 (21.796) | 33.39 (30.847) | 43.88 (32.419)

8. Secondary Outcome: Total Consumption of Rescue Medication
Description: The total consumption of rescue analgesia was reported.
Time Frame: 7 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: oral morphine equivalents
Arm/Group | PGB and APAP (Group A) | APAP (Group B) | Placebo (Group C).
Number analyzed (Participants) | 35 | 35 | 17
oral morphine equivalents | 17.79 (22.344) | 34.24 (32.496) | 44.76 (33.609)

9. Secondary Outcome: Time to First Use of Rescue Medication From Hour 0
Description: Time to first use of rescue medication from Hour 0 was reported. Hour 0 was defined as the end of surgery (i.e., completion of the last suture).
Time Frame: 7 days
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: hours
Arm/Group | PGB and APAP (Group A) | APAP (Group B) | Placebo (Group C).
Number analyzed (Participants) | 20 | 28 | 14
hours | 11.60 [5.93 to 16.12] | 5.78 [4.27 to 7.97] | 4.31 [3.57 to 5.87]

10. Secondary Outcome: Percentage of Participants Who Used Rescue Medication
Description: Percentage of participants who used rescue medication is reported
Time Frame: 7 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | PGB and APAP (Group A) | APAP (Group B) | Placebo (Group C).
Number analyzed (Participants) | 35 | 35 | 17
percentage of participants | 57.1 | 80.0 | 82.4

11. Secondary Outcome: Patient Global Assessment of Pain
Description: Patient Global Assessment (PGA) of pain control at 48 hours was reported. Patient global evaluation will be self-reported over 24 hours, using a 0-4 categorical rating scale of: (0) poor, (1) fair, (2) good, (3) very good, and (4) excellent
Time Frame: 48 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PGB and APAP (Group A) | APAP (Group B) | Placebo (Group C).
Number analyzed (Participants) | 35 | 34 | 15
Participants
  (0) Poor | 1 | 1 | 1
  (1) Fair | 4 | 7 | 7
  (2) Good | 6 | 7 | 3
  (3) Very good | 10 | 10 | 3
  (4) Excellent | 14 | 9 | 1

12. Secondary Outcome: Maximum Observed Concentration for PGB and APAP
Description: The Plasma Concentration (Cmax) is defined as the maximum observed concentration. Multiple blood samples were drawn at pre-decided time points. Timing for blood draws was within 3 minutes of the end of every infusion. Three minutes was the maximum allowance as every effort was made to take the sample as close as possible to 1.0 minute after infusion.
Time Frame: Pre-infusion (at least 3.0 minutes before the start of the first infusion) and at 0.5, 1.5, 6.0, 8.0, 12.0, 16.0, 18.0, 24.0, 30.0, 32.0, 36.0, 40.0, 42.0, and 48 hours post-infusion
Population: The PK Analysis Set included all randomized subjects who received any amount of study drug, had no protocol deviations affecting the pharmacokinetic (PK) variables, and had sufficient data collected to allow evaluation of least one PK parameter (minimum plasma concentration of the drug [Cmin], Cmax, or both). Subjects were analyzed according to treatment received. All PK analyses were performed using the PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/ml)
Arm/Group | PGB and APAP (Group A) | APAP (Group B) | Placebo (Group C).
Number analyzed (Participants) | 34 | 33 | 0
nanogram per milliliter (ng/ml)
  Mean Cmax Values of Pregabalin- First Dose: number analyzed (Participants) | 33 | 0 | 0
  Mean Cmax Values of Pregabalin- First Dose | 10068 (36) |  |
  Mean Cmax Values of Pregabalin- Last Dose: number analyzed (Participants) | 33 | 0 | 0
  Mean Cmax Values of Pregabalin- Last Dose | 12960 (27) |  |
  Mean Cmax Values of Acetaminophen-First Dose: number analyzed (Participants) | 33 | 33 | 0
  Mean Cmax Values of Acetaminophen-First Dose | 28700 (34) | 16847 (39) |

13. Secondary Outcome: Minimum Observed Concentration for PGB and APAP
Description: The Plasma Concentration (Cmin) is defined as the minimum observed concentration. Multiple blood samples were drawn at pre-decided time points. Timing for blood draws was within 3 minutes of the end of every infusion. Three minutes was the maximum allowance as every effort was made to take the sample as close as possible to 1.0 minute after infusion.
Time Frame: as for outcome 12
Population: The PK Analysis Set included all randomized subjects who received any amount of study drug, had no protocol deviations affecting the PK variables, and had sufficient data collected to allow evaluation of least one PK parameter (minimum plasma concentration of the drug [Cmin], Cmax, or both). Subjects were analyzed according to treatment received. All PK analyses were performed using the PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/ml)
Arm/Group | PGB and APAP (Group A) | APAP (Group B) | Placebo (Group C).
Number analyzed (Participants) | 34 | 33 | 0
nanogram per milliliter (ng/ml) | NA (NA) — Aside from the pre-dose sample collected just before the start of the first dose, there were no samples taken prior to each dose. Therefore, Cmin was unable to be estimated from the available samples. | NA (NA) — Aside from the pre-dose sample collected just before the start of the first dose, there were no samples taken prior to each dose. Therefore, Cmin was unable to be estimated from the available samples. |

ADVERSE EVENTS:
Time Frame: Up to 7 days (± 1 day)
Description: An adverse event (AE) is defined as any untoward medical occurrence and does not necessarily have to have causal relationship with the study medication. An AE can therefore be an unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease, which is a change from baseline and is temporally associated with the use of the study medication, whether or not it is considered related to the study medication.
Arm/Group | PGB and APAP (Group A) | APAP (Group B) | Placebo (Group C).
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/17
Other Adverse Events (participants affected / at risk) | 27/35 | 15/35 | 9/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PGB and APAP (Group A) (N=35) | APAP (Group B) (N=35) | Placebo (Group C). (N=17)
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Diplopia (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 9 | 5 | 5
Vomiting (Gastrointestinal disorders) | 5 | 2 | 4
Application site rash (General disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 1 | 0
Infusion site extravasation (General disorders) | 1 | 0 | 0
Injection site erythema (General disorders) | 1 | 0 | 0
Injection site extravasation (General disorders) | 2 | 0 | 1
Pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0
Post procedural cellulitis (Infections and infestations) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Transaminases abnormal (Investigations) | 1 | 0 | 0
Transaminases increased (Investigations) | 2 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 18 | 3 | 3
Headache (Nervous system disorders) | 3 | 2 | 2
Presyncope (Nervous system disorders) | 1 | 0 | 0
Euphoric mood (Psychiatric disorders) | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/83/NCT04495283/Prot_SAP_000.pdf